CLINICAL TRIAL: NCT06048887
Title: A Double-blind, Randomized, Placebo-controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of CRN04894 in Healthy Volunteers
Brief Title: Single and Multiple-Ascending Dose Study of CRN04894 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Crinetics Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRN04894-01
Record Dates: First submitted 2023-09-11; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single Ascending Dose (Part 1) (Experimental)
  Interventions: Drug: CRN04894 Oral Solution; Drug: Placebo Oral Solution
- Multiple Ascending Dose (Part 2) (Experimental)
  Interventions: Drug: CRN04894 Oral Solution; Drug: Placebo Oral Solution

INTERVENTIONS:
Drug: CRN04894 Oral Solution — CRN04894 is an orally active nonpeptide melanocortin 2 receptor (MC2R) or adrenocorticotropic hormone (ACTH) antagonist.
Drug: Placebo Oral Solution — Placebo

SUMMARY:
A Phase 1, first-in-human, double-blind, randomized, placebo-controlled study to evaluate the safety of CRN04894 in healthy volunteers as well as the relationship between exposure and pharmacodynamic (PD) parameters.

ELIGIBILITY:
Inclusion Criteria:

* Females must be either postmenopausal or surgically sterile; or using stable and permitted highly effective method of contraception - use of oral hormonal contraceptives are not allowed during the study
* Male subjects must be surgically sterile or agree to use highly effective form of contraception when sexually active with a female partner of child bearing potential
* ACTH-stimulated serum cortisol high-dose ACTH stimulation test conducted at Screening

Exclusion Criteria:

* Use of topical, nasal, inhaled, or oral corticosteroids.
* Use of any investigational drug within the past 60 days.
* Have a medically significant illness within 30 days prior to screening.
* Use of prohibited prescribed or nonprescribed medications and/or nonmedications/alternative medicinal products.
* Any condition that in the opinion of the investigator would jeopardize the subject's appropriate participation in this study.
* Unstable psychological disorder ≤1 year prior to Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with treatment-emergent adverse events | Part 1 - up to Day 8; Part 2 - up to Day 20
Proportion of participants with a clinically significant safety laboratory observation | Part 1 - up to Day 8; Part 2 - up to Day 20

SECONDARY OUTCOMES:
Pharmacokinetics (AUC) | Part 1 - up to Day 8; Part 2 - up to Day 20
  Assessment of the plasma area under the curve of CRN04894
Pharmacokinetics (Cmax) | Part 1 - up to Day 8; Part 2 - up to Day 20
  Assessment of the maximum observed plasma concentration of CRN04894
Pharmacokinetics (Tmax) | Part 1 - up to Day 8; Part 2 - up to Day 20
  Assessment of time to maximal CRN04894 concentration (Tmax)
Pharmacokinetics (T1/2) | Part 1 - up to Day 8; Part 2 - up to Day 20
  Assessment of elimination half-life of CRN04894

OTHER OUTCOMES:
Change in ACTH-stimulated serum cortisol | Part 1 - Day 1; Part 2 - Day 10
Change in serum cortisol | Part 1 - up to Day 8; Part 2 - up to Day 20

CONTACTS AND LOCATIONS:
Locations (1):
- QPS-Miami Research Associates, Miami, Florida, United States